CLINICAL TRIAL: NCT00481182
Title: A Phase I, Open-Label, 2-Period, Single-Sequence, Drug Interaction Study to Assess Steady-State Plasma Methadone Enantiomer Pharmacokinetics Following Co-Administration of Methadone QD With Fosamprenavir 700mg BID + RTV 100mg BID in Opiate-Dependent, HIV Seronegative, Adult Subjects
Brief Title: Co-Administration Of Fosamprenavir With Methadone: A Drug Interaction Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102577
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2009-02-23 (Estimated); Status verified 2009-02

CONDITIONS: Healthy Subjects
Keywords: PK; PD; FPV; RTV; APV; ritonavir; fosamprenavir; amprenavir; methadone; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — fosamprenavir; Ritonavir; Methadone

INTERVENTIONS:
Drug: fosamprenavir + ritonavir + methadone

SUMMARY:
To assess the combined effects of fosamprenavir 700mg BID + ritonavir 100mg BID + standardized dose of methadone, on plasma total and unbound methadone enantiomer pharmacokinetics (PK), opiate pharmacodynamic (PD) measures, and safety. The effect of methadone on plasma amprenavir PK will also be assessed by comparison to historical control data.

ELIGIBILITY:
Inclusion Criteria:

* Subject is enrolled in a certified methadone maintenance program for at least 12 weeks prior to Period 1, Day 1.

Subject is receiving methadone = 200mg QD that has remained unchanged for 30 days The subject is male, female and is between the age of 18 and 64 years of age.

A female is eligible to enter and participate if she is of non-childbearing potential or of childbearing potential. If of childbearing potential, females must have a negative serum pregnancy test at Screening, and agree to one of the following:

Complete abstinence from sexual intercourse from 2 weeks prior to administration of the study drug. Sexual intercourse with only vasectomized partner.

Body mass index of 19.00 to 32.00 kg/m2. Willing to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.

Able to understand and comply with protocol requirements and instructions and is likely to complete the study as planned.

Able to give written informed consent prior to screening.

Exclusion Criteria:

* Subject has a clinically significant abnormality identified on the screening medical or laboratory evaluation, including 12-lead ECG.

Subject has any preexisting condition which could interfere with the absorption, metabolism, and/or excretion of the study drugs.

Subject currently has or has a history of decompensated liver disease (i.e., ascites, esophageal or rectal varices, hepatic encephalopathy) or current evidence of active hepatitis (AST or ALT > 2.5x ULN).

Subject has evidence of liver impairment at screening (i.e., INR > 1.7, total bilirubin >2.0 mg/dL, albumin <3.5 g/dL).

Subject has inadequate venous access. Subject has a history of any hypersensitivity reaction to any component of FPV, APV, RTV, or to any drug chemically related to FPV, APV, or RTV.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-02

PRIMARY OUTCOMES:
Serial blood samples will be collected over 24 hours for measurement of plasma (R-) and (S-) methadone (days 4 and 18) and serum amprenavir concentrations (day 18).

SECONDARY OUTCOMES:
On study days 4, 11, and 18, opioid effects will be assessed pre-dose, 2 hours, and 6 hours following methadone dosing. Pharmacokinetic and opioid pharmacodynamic parameters will be compared between the two treatments.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Buffalo, New York